CLINICAL TRIAL: NCT06085209
Title: Cryospray Therapy for Benign Airway Stenosis: a Pilot Study (Pilot-CRYOSTASIS)
Brief Title: Cryospray Therapy for Benign Airway Stenosis
Acronym: CRYOSTASIS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: US Endoscopy Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20027230
Record Dates: First submitted 2023-09-28; First posted 2023-10-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Stenosis Trachea
Keywords: cryospray therapy; benign airway stenosis
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a 1:1 fashion to intervention standard of care (SOC) + SCT and control (SOC) groups. Participants will be blinded to the use of SCT to prevent knowledge of their group assignment from biasing their subjective assessments. Adjudicators in the primary outcome measurements (quantitative CT) will be blinded to group assignment as well.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the use of SCT to prevent knowledge of their group assignment from biasing their subjective assessments. Adjudicators in the primary outcome measurements (quantitative CT) will be blinded to group assignment as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Bronchoscopic balloon dilation with radial cuts & truFreeze spray cryotherapy
  Interventions: Device: The truFreeze Spray Cryotherapy; Device: Ballon dilation; Device: Radial Incision
- Standard of care (Active Comparator): Bronchoscopic balloon dilation with radial cuts
  Interventions: Device: Ballon dilation; Device: Radial Incision

INTERVENTIONS:
Device: The truFreeze Spray Cryotherapy — A novel FDA cleared technique that allows for liquid nitrogen (LN2) to be delivered in a metered fashion via a catheter through a flexible bronchoscope.
  Arms: Intervention
Device: Ballon dilation — An endoscopic balloon that is inflated with water to pressures between 45 and 131 psi (3-9 atm) using a syringe and pressure manometer.
Device: Radial Incision — Carbon dioxide (CO2) laser or Monopolar electrocautery knife

SUMMARY:
This is a clinical evaluation to assess the effectiveness of cryospray therapy used in addition to current standard of care endoscopic therapies in preventing short term recurrent airway stenosis with a multicentric outcome evaluation. The investigators hypothesize that the addition of SCT to standard endoscopic treatment of benign airway stenosis will result in decreased stenosis recurrence at 6 months as estimated by quantitative radiologic assessment of the stenotic volume.

DETAILED DESCRIPTION:
Spray cryo treatment of tracheal stenosis has the potential for long-lasting endoscopic management of BCAS and is used as part of routine clinical care by many physicians, but there is a relative paucity of peer-reviewed data, and no randomized controlled trial has been performed. Thus, the study could potentially show that the use of spray cryo therapy could allow patients to undergo fewer procedures to treat this condition, or lengthen the amount of time required in between these procedures, or play a role in the resolution of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Referral to interventional pulmonology or otorhinolaryngology or thoracic surgery for endoscopic management of suspected benign tracheal stenosis.
* Significant tracheal stenosis defined by stenosis ≥ 50% of tracheal lumen assessed on chest CT or previous bronchoscopy
* Able to provide informed consent.
* Age > 18

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Known or suspected malignant central airway stenosis
* Patient has already been enrolled in this study.
* Study subject has any disease or condition that interferes with safe completion of the study including:

  1. Hypoxemia with need for supplemental oxygen ≥ 2L/min by nasal canula
  2. Pneumothorax in the previous 12 months
  3. Severe COPD (defined as a FEV1/FVC < 70% and FEV1 <30% predicted) and/or severe persistent asthma.
  4. Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the attending physicians.
  5. Compromised tissue where significant ulceration or mucosal break is evident in the ablation area or adjacent organs.
  6. Significantly reduced tissue strength caused by prior procedure or pre-existing condition (e.g. PEG tube)
  7. Significantly reduced elasticity of the ablation area (e.g. Marfan's Syndrome)
* Prior complications with SCT (Spray cryotherapy)
* Contraindication to rigid bronchoscopy
* Significant tracheomalacia or alterations in cartilage integrity on CT (Computed Tomography) that would require stent placement or surgical referral.
* Greater than 1 BCAS intervention, excluding cricotracheal (tracheal surgery) resection, within 6 months before enrollment.
* Anatomical flow resistance (gas evacuation) where any procedure or anatomy proximal to the ablation site has significantly reduced or restricted the flow area of the lumen creating restriction where gas created from liquid nitrogen cannot adequately vent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Degree of re-stenosis | 6 months
  The degree of re-stenosis at 6 months expressed as the percentage of airway lumen volume within the stenotic segment at 6 months compared to personal best patency volume on CT scan performed within five weeks of the study intervention.

SECONDARY OUTCOMES:
Change in Peak Expiratory Flow (PEF) | Continous for 6 months
  Evidence supports the use of PEF as a simple, efficient, and accessible way of monitoring progression of tracheal stenosis. PEF has previously been captured in clinical encounters as component of the decision-making algorithm for surgical intervention in tracheal stenosis patients. Mobile Device Software 'App' can robustly capture longitudinal patient reported outcome measures. A previously developed mobile device software 'Airflo' for tracking patient-generated health data and has proven the ability to successfully implement this software.
Clinical Chronic Obstructive Pulmonary Disease Questionnaire (CCQ) | 2 weeks before procedure, 2 weeks after the procedure, the 3 month study mark, the 6 months study mark,
  The CCQ has been used as a validated quality of life measure in laryngotracheal stenosis. The investigators will send surveys out to patients at set time intervals to assess symptom improvement pre- and post-intervention. The questions are divided into three areas or domains. Symptoms 1, 2, 5, 6; Functional state 7, 8, 9, 10; Mental state 3 and 4. All items are equally weighted by adding score of ten items and dividing by the number ten. The score varies between 0 (very good health status) to 6 (extremely poor health status).
Incidence of complications between groups | Continous for 6 months
  Incidence of complications (hypoxemia, bleeding, pneumothorax rate, barotrauma).

CONTACTS AND LOCATIONS:
Overall Officials: Ray Shepherd, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virgnia Commonwealth University, Richmond, Virginia, United States